CLINICAL TRIAL: NCT06069206
Title: Effect of Direct-from-blood Bacterial Testing on Antibiotic Administration and Clinical Outcomes: A Learning Healthcare Pragmatic Randomized Trial
Brief Title: Effect of Direct-from-blood Bacterial Testing on Antibiotic Administration and Clinical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Semler, MD, MSc, Medical Director, Center for Learning Healthcare; Associate Director, Vanderbilt Medical Intensive Care Unit, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 231229
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Bloodstream Infection; Sepsis Bacterial; MRSA Bacteremia; Vancomycin
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: This study will be performed as a pragmatic, randomized controlled clinical trial with parallel group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Patients will receive blood cultures and will not receive direct-from-blood testing.
  Interventions: Other: Usual Care
- Direct-from-blood testing (Active Comparator): In addition to usual care, patients will receive direct-from-blood testing using the T2Bacteria® Panel.
  Interventions: Other: T2Bacteria® Panel (direct-from-blood testing)

INTERVENTIONS:
Other: T2Bacteria® Panel (direct-from-blood testing) — Providers will be prompted to order the T2Bacteria® Panel (direct-from-blood testing) and accompanying communications regarding panel results will be delivered.
  Arms: Direct-from-blood testing
Other: Usual Care — Standard blood cultures.
  Arms: Usual Care

SUMMARY:
Bacterial blood stream infections are common and life-threatening. Bloodstream infections have historically been identified using blood cultures, which often take 24-72 hours to result and are imperfectly sensitive. Early administration of antimicrobial therapy is a fundamental component of the management of adults presenting to the hospital with a suspected bloodstream infection and/or sepsis.

But because blood cultures frequently take 24-72 hours to result, patients are typically treated with empiric, broad spectrum antibiotics. In a meta-analysis of sepsis studies, empirical antibiotic therapy was inappropriate for the organism that ultimately grew in culture in almost half of patients. Thus, patients are commonly exposed to unnecessary antibiotics without evidence of infection or with evidence of infection requiring narrow antibiotic selection. For example, current guidelines recommend the use of empiric intravenous vancomycin as coverage for a bloodstream infection caused by the bacterial pathogen methicillin-resistant S. aureus (MRSA). Vancomycin requires careful monitoring due to its narrow therapeutic range and high risk of toxicity. Administration of vancomycin to patients who do not have MRSA can lead to avoidable adverse drug events and costs, as well as drive antimicrobial resistance.

There has been increasing interest in using rapid diagnostic tests that identify bacteria directly from whole blood samples without relying on growth in culture, referred to as "direct-from-blood" tests, to guide early therapeutic management of patients with suspected bloodstream infections in addition to standard blood cultures. One such FDA-approved, direct-from-blood test is the T2Bacteria® Panel. This panel's performance as a direct-from blood test for bacterial pathogens has been described in previous studies. A recent meta-analysis of largely observational studies reported a faster transition to targeted microbial therapy and de-escalation of empirical microbial therapy, as well as a shorter duration of intensive care unit stay and hospital stay for patients who received this direct-from-blood test.

We will conduct a pragmatic, randomized clinical trial examining the effect of using the T2Bacteria® Panel direct from-blood testing, compared to using blood cultures alone (standard of care), on antimicrobial receipt and clinical outcomes for adults presenting to the hospital with suspected infection and who have been initiated on empiric therapy with intravenous vancomycin.

ELIGIBILITY:
Inclusion Criteria:

* Patient is located in the Emergency Department at Vanderbilt University Hospital
* ≤ 12 hours from patient presentation to the Emergency Department at Vanderbilt University Hospital
* Age ≥ 18 years
* Clinician has ordered blood cultures
* Clinician has ordered intravenous vancomycin

Exclusion Criteria:

* Patient is known to be a prisoner
* Patient is known to be pregnant
* Patient is known to have received 2 or more doses of vancomycin since presentation to the Vanderbilt ED
* Patient is known to have a positive bacterial culture in the previous 7 days
* Patient is known to have an infection for which at least 7 days of intravenous vancomycin would routinely be administered regardless of bacterial testing results (e.g., skin and soft tissue infection, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Time to last dose of intravenous vancomycin | Baseline to 14 days
  The time between randomization and the start time for the last dose of intravenous vancomycin received by the patient within 14 days of randomization.

SECONDARY OUTCOMES:
Time to last dose of systemic anti-pseudomonal beta-lactam antibiotic | Baseline to 14 days
  The time between randomization and start time of the last dose of systemic anti-pseudomonal beta-lactam antibiotic received by the patient within 14 days of randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Semler, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Background] Opota O, Croxatto A, Prod'hom G, Greub G. Blood culture-based diagnosis of bacteraemia: state of the art. Clin Microbiol Infect. 2015 Apr;21(4):313-22. doi: 10.1016/j.cmi.2015.01.003. Epub 2015 Jan 16. PMID 25753137
- [Background] Leggieri N, Rida A, Francois P, Schrenzel J. Molecular diagnosis of bloodstream infections: planning to (physically) reach the bedside. Curr Opin Infect Dis. 2010 Aug;23(4):311-9. doi: 10.1097/QCO.0b013e32833bfc44. PMID 20592531
- [Background] Shah SS, Downes KJ, Elliott MR, Bell LM, McGowan KL, Metlay JP. How long does it take to "rule out" bacteremia in children with central venous catheters? Pediatrics. 2008 Jan;121(1):135-41. doi: 10.1542/peds.2007-1387. PMID 18166567
- [Background] Peralta G, Rodriguez-Lera MJ, Garrido JC, Ansorena L, Roiz MP. Time to positivity in blood cultures of adults with Streptococcus pneumoniae bacteremia. BMC Infect Dis. 2006 Apr 27;6:79. doi: 10.1186/1471-2334-6-79. PMID 16643662
- [Background] Tabak YP, Vankeepuram L, Ye G, Jeffers K, Gupta V, Murray PR. Blood Culture Turnaround Time in U.S. Acute Care Hospitals and Implications for Laboratory Process Optimization. J Clin Microbiol. 2018 Nov 27;56(12):e00500-18. doi: 10.1128/JCM.00500-18. Print 2018 Dec. PMID 30135230
- [Background] Paul M, Shani V, Muchtar E, Kariv G, Robenshtok E, Leibovici L. Systematic review and meta-analysis of the efficacy of appropriate empiric antibiotic therapy for sepsis. Antimicrob Agents Chemother. 2010 Nov;54(11):4851-63. doi: 10.1128/AAC.00627-10. Epub 2010 Aug 23. PMID 20733044
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children: executive summary. Clin Infect Dis. 2011 Feb 1;52(3):285-92. doi: 10.1093/cid/cir034. PMID 21217178
- [Background] Rybak MJ, Le J, Lodise TP, Levine DP, Bradley JS, Liu C, Mueller BA, Pai MP, Wong-Beringer A, Rotschafer JC, Rodvold KA, Maples HD, Lomaestro BM. Therapeutic monitoring of vancomycin for serious methicillin-resistant Staphylococcus aureus infections: A revised consensus guideline and review by the American Society of Health-System Pharmacists, the Infectious Diseases Society of America, the Pediatric Infectious Diseases Society, and the Society of Infectious Diseases Pharmacists. Am J Health Syst Pharm. 2020 May 19;77(11):835-864. doi: 10.1093/ajhp/zxaa036. No abstract available. PMID 32191793
- [Background] Peri AM, Stewart A, Hume A, Irwin A, Harris PNA. New Microbiological Techniques for the Diagnosis of Bacterial Infections and Sepsis in ICU Including Point of Care. Curr Infect Dis Rep. 2021;23(8):12. doi: 10.1007/s11908-021-00755-0. Epub 2021 Jun 16. PMID 34149321
- [Background] Timbrook TT, Morton JB, McConeghy KW, Caffrey AR, Mylonakis E, LaPlante KL. The Effect of Molecular Rapid Diagnostic Testing on Clinical Outcomes in Bloodstream Infections: A Systematic Review and Meta-analysis. Clin Infect Dis. 2017 Jan 1;64(1):15-23. doi: 10.1093/cid/ciw649. Epub 2016 Sep 26. PMID 27678085
- [Background] Pliakos EE, Andreatos N, Shehadeh F, Ziakas PD, Mylonakis E. The Cost-Effectiveness of Rapid Diagnostic Testing for the Diagnosis of Bloodstream Infections with or without Antimicrobial Stewardship. Clin Microbiol Rev. 2018 May 30;31(3):e00095-17. doi: 10.1128/CMR.00095-17. Print 2018 Jul. PMID 29848775
- [Background] Nguyen MH, Clancy CJ, Pasculle AW, Pappas PG, Alangaden G, Pankey GA, Schmitt BH, Rasool A, Weinstein MP, Widen R, Hernandez DR, Wolk DM, Walsh TJ, Perfect JR, Wilson MN, Mylonakis E. Performance of the T2Bacteria Panel for Diagnosing Bloodstream Infections: A Diagnostic Accuracy Study. Ann Intern Med. 2019 Jun 18;170(12):845-852. doi: 10.7326/M18-2772. Epub 2019 May 14. PMID 31083728
- [Background] Voigt C, Silbert S, Widen RH, Marturano JE, Lowery TJ, Ashcraft D, Pankey G. The T2Bacteria Assay Is a Sensitive and Rapid Detector of Bacteremia That Can Be Initiated in the Emergency Department and Has Potential to Favorably Influence Subsequent Therapy. J Emerg Med. 2020 May;58(5):785-796. doi: 10.1016/j.jemermed.2019.11.028. Epub 2020 Jan 23. PMID 31982197
- [Background] Drevinek P, Hurych J, Antuskova M, Tkadlec J, Berousek J, Prikrylova Z, Bures J, Vajter J, Soucek M, Masopust J, Martinkova V, Adamkova J, Hysperska V, Bebrova E. Direct detection of ESKAPEc pathogens from whole blood using the T2Bacteria Panel allows early antimicrobial stewardship intervention in patients with sepsis. Microbiologyopen. 2021 Jun;10(3):e1210. doi: 10.1002/mbo3.1210. PMID 34180598
- [Background] De Angelis G, Posteraro B, De Carolis E, Menchinelli G, Franceschi F, Tumbarello M, De Pascale G, Spanu T, Sanguinetti M. T2Bacteria magnetic resonance assay for the rapid detection of ESKAPEc pathogens directly in whole blood. J Antimicrob Chemother. 2018 Mar 1;73(suppl_4):iv20-iv26. doi: 10.1093/jac/dky049. PMID 29608753
- [Background] Giannella M, Pankey GA, Pascale R, Miller VM, Miller LE, Seitz T. Antimicrobial and resource utilization with T2 magnetic resonance for rapid diagnosis of bloodstream infections: systematic review with meta-analysis of controlled studies. Expert Rev Med Devices. 2021 May;18(5):473-482. doi: 10.1080/17434440.2021.1919508. Epub 2021 Jun 7. PMID 33863237
- [Derived] Gaston DC, Humphries RM, Lewis AA, Gatto CL, Wang L, Nelson GE, Stollings JL, Ereshefsky BJ, Christensen MA, Dear ML, Banerjee R, Miller KF, Self WH, Semler MW, Qian ET; Vanderbilt Center for Learning Healthcare. Examining the effect of direct-from-blood bacterial testing on antibiotic administration and clinical outcomes: a protocol and statistical analysis plan for a pragmatic randomised trial. BMJ Open. 2025 Jan 11;15(1):e090263. doi: 10.1136/bmjopen-2024-090263. PMID 39800394